CLINICAL TRIAL: NCT03401788
Title: An Open-Label Phase 2 Study to Evaluate PT2977 for the Treatment of Von Hippel Lindau Disease-Associated Renal Cell Carcinoma
Brief Title: A Phase 2 Study of Belzutifan (PT2977, MK-6482) for the Treatment of Von Hippel Lindau (VHL) Disease-Associated Renal Cell Carcinoma (RCC) (MK-6482-004)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peloton Therapeutics, Inc., a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6482-004; PT2977-202 (Other: Peloton Study ID); MK-6482-004 (Other: MSD); 2023-509119-99 (Registry Identifier: EU CT Number); 2018-000125-30 (EudraCT Number)
Record Dates: First submitted 2018-01-09; First posted 2018-01-17 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: VHL - Von Hippel-Lindau Syndrome; VHL Gene Mutation; VHL Syndrome; VHL Gene Inactivation; VHL-Associated Renal Cell Carcinoma; VHL-Associated Clear Cell Renal Cell Carcinoma
Keywords: VHL
MeSH Terms: conditions — von Hippel-Lindau Disease | interventions — belzutifan

STUDY DESIGN:
Intervention Model Description: Phase 2 Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open Label Belzutifan (Experimental): Participants receive 120 mg belzutifan orally once daily. Participants may continue to receive belzutifan in the absence of unacceptable treatment related toxicity or unequivocal disease progression.
  Interventions: Drug: Belzutifan

INTERVENTIONS:
Drug: Belzutifan — 120 mg once daily (three 40 mg oral tablets once daily).
  Other Names: PT2977; MK-6482; WELIREG™

SUMMARY:
This study is designed to investigate belzutifan as a treatment for VHL disease associated RCC.

DETAILED DESCRIPTION:
This open-label Phase 2 study will evaluate the efficacy and safety of belzutifan in participants with VHL disease who have at least 1 measurable RCC tumor. Belzutifan will be administered orally and treatment will be continuous. Participants will be evaluated radiologically approximately 12 weeks after initiation of treatment and every 12 weeks thereafter while continuing in the study for a minimum of 3 years and then every 24 weeks or more frequently if clinically indicated. Changes in VHL disease-associated non-RCC tumors will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Has a diagnosis of von Hippel Lindau disease, based on a germline VHL alteration
* Has at least 1 measurable solid RCC tumor and no RCC tumor that requires immediate surgical intervention. The diagnosis of RCC can be radiologic (histologic diagnosis not required). Participants may have VHL disease-associated tumors in other organ systems

Exclusion Criteria:

* Has received prior treatment with belzutifan or another HIF-2α inhibitor
* Has had any systemic anti-cancer therapy (includes anti-vascular endothelial growth factor [VEGF] therapy or any systemic investigational anti-cancer agent)
* Has an immediate need for surgical intervention for tumor treatment
* Has evidence of metastatic disease on screening imaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-05-02 (Actual); Primary Completion 2026-03-29 (Estimated); Study Completion 2026-03-29 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) in VHL Disease-Associated RCC Tumors | Up to approximately 4 years
  ORR is defined as the percentage of participants in the analysis population who have a best confirmed response of Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1). ORR will be assessed by independent review committee (ICR) for the primary analysis.

SECONDARY OUTCOMES:
Duration of Response (DOR) in VHL Disease-Associated RCC Tumors | Up to approximately 4 years
  DOR is defined as the interval from the first documented evidence of a CR (disappearance of all target lesions) or a PR (at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1 until Progressive Disease (PD) or death due to any cause, whichever occurs first, in participants demonstrating a best confirmed response of CR or PR. Per RECIST 1.1, PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD.
Time to Response (TTR) in VHL Disease-Associated RCC Tumors | Up to approximately 4 years
  TTR is defined as the interval from the start of study treatment to the first documentation of a response per RECIST 1.1, and calculated for participants with a best confirmed response of CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions).
Progression-free Survival (PFS) in VHL Disease-Associated RCC Tumors | Up to approximately 4 years
  PFS is defined as the interval from the start of study treatment to the first documented PD or death from any cause, whichever occurs first. Per RECIST 1.1, PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD.
Time to Surgery (TTS) in VHL Disease-Associated RCC Tumors | Up to approximately 4 years
  TTS was defined as the interval from the start of study treatment to the date of surgery.
ORR in VHL Disease-Associated Non-RCC Tumors | Up to approximately 4 years
  ORR is defined as the percentage of participants in the analysis population who have a best confirmed response of CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1.
DOR in VHL Disease-Associated Non-RCC Tumors | Up to approximately 4 years
  DOR is defined as the interval from the first documented evidence of a CR (disappearance of all target lesions) or a PR (at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1 until PD or death due to any cause, whichever occurs first, in participants demonstrating a best confirmed response of CR or PR. Per RECIST 1.1, PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD.
TTR in VHL Disease-Associated Non-RCC Tumors | Up to approximately 4 years
  TTR is defined as the interval from the start of study treatment to the first documentation of a response per RECIST 1.1, and calculated for participants with a best confirmed response of CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions).
PFS in VHL Disease-Associated Non-RCC Tumors | Up to approximately 4 years
  PFS is defined as the interval from the start of study treatment to the first documented PD or death from any cause, whichever occurs first. Per RECIST 1.1, PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD.
TTS in VHL Disease-Associated Non-RCC Tumors | Up to approximately 4 years
  TTS was defined as the interval from the start of study treatment to the date of surgery.
Number of Participants Experiencing an Adverse Event (AE) | Up to approximately 4 years
  An AE is any untoward medical occurrence in a participant regardless of its causal relationship to study treatment. An AE can be any unfavorable and unintended sign (including any clinically significant abnormal laboratory test result), symptom, or disease temporally associated with the use of the study drug, whether or not it is considered to be study drug related.
Number of Participants Experiencing a Serious Adverse Event (SAE) | Up to approximately 4 years
  An SAE is any AE occurring at any dose and regardless of causality that meets any of the following criteria: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, is a congenital anomaly or birth defect in an offspring of a participant taking study drug, or is an important medical event.
Belzutifan Plasma Concentration | Weeks 1 and 3: pre-dose, 2 and 5 hours post-dose, Week 5, 9, and 13: post-dose.
  Blood samples for the determination of belzutifan concentration will be collected at pre-specified timepoints before and after treatment administration.
Belzutifan Metabolite Plasma Concentration | Weeks 1 and 3: pre-dose, 2 and 5 hours post-dose, Week 5, 9, and 13: post-dose.
  Blood samples for the determination of belzutifan metabolite concentration will be collected at pre-specified timepoints before and after treatment administration.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (11):
- United States (8):
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - University of Pennsylvania Medical Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Vanderbilt Medical Center, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
- Aarhus University Hospital, Aarhus, Denmark
- Hospital Georges Pompidou, Paris, France
- Cambridge University Hospital, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Iliopoulos O, Iversen AB, Narayan V, Maughan BL, Beckermann KE, Oudard S, Else T, Maranchie JK, Goldberg CM, Fu W, Perini RF, Liu Y, Linehan WM, Srinivasan R, Jonasch E. Belzutifan for patients with von Hippel-Lindau disease-associated CNS haemangioblastomas (LITESPARK-004): a multicentre, single-arm, phase 2 study. Lancet Oncol. 2024 Oct;25(10):1325-1336. doi: 10.1016/S1470-2045(24)00389-9. Epub 2024 Sep 13. PMID 39284337
- [Derived] Srinivasan R, Iliopoulos O, Beckermann KE, Narayan V, Maughan BL, Oudard S, Else T, Maranchie JK, Iversen AB, Cornell J, Perini RF, Liu Y, Linehan WM, Jonasch E. Belzutifan for von Hippel-Lindau disease-associated renal cell carcinoma and other neoplasms (LITESPARK-004): 50 months follow-up from a single-arm, phase 2 study. Lancet Oncol. 2025 May;26(5):571-582. doi: 10.1016/S1470-2045(25)00099-3. Epub 2025 Apr 12. PMID 40228516
- [Derived] Jonasch E, Donskov F, Iliopoulos O, Rathmell WK, Narayan VK, Maughan BL, Oudard S, Else T, Maranchie JK, Welsh SJ, Thamake S, Park EK, Perini RF, Linehan WM, Srinivasan R; MK-6482-004 Investigators. Belzutifan for Renal Cell Carcinoma in von Hippel-Lindau Disease. N Engl J Med. 2021 Nov 25;385(22):2036-2046. doi: 10.1056/NEJMoa2103425. PMID 34818478
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26345&tenant=MT_MSD_9011